CLINICAL TRIAL: NCT02832063
Title: A Randomized, Double Blinded, Phase IIb/III, Decentralized Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Participants With Mild to Moderate Acne Vulgaris
Brief Title: Clinical Trial in Subjects With Mild to Moderate Acne Vulgaris
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AOBiome LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVB244-002
Record Dates: First submitted 2016-07-08; First posted 2016-07-13 (Estimated); Results first posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- B244 arm (Active Comparator): B244 dose administered in a 1:1 (active vs placebo) ratio
  Interventions: Biological: B244
- Placebo arm (Placebo Comparator): Placebo dose administered in a 1:1 (active vs placebo) ratio
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: B244 — 4 pumps of spray to saturate the entire face applied BID. Applications should occur in the morning and at night for 12 weeks.
  Arms: B244 arm
Biological: Placebo — 4 pumps of spray to saturate the entire face applied BID. Applications should occur in the morning and at night for 12 weeks.
  Arms: Placebo arm

SUMMARY:
The purpose of this study is to demonstrate the safety, tolerability and efficacy of B244 administered over 12 weeks to participants with mild to moderate acne vulgaris relative to placebo.

DETAILED DESCRIPTION:
This is a Phase IIb/III, randomized, double blinded, decentralized clinical trial evaluating the safety, tolerability, and efficacy of B244 compared to placebo in the treatment of acne vulgaris

1.1. Primary Objectives

1. To evaluate the safety and tolerability of B244 in participants with acne vulgaris
2. To assess the efficacy of B244 in participants with mild to moderate acne vulgaris from baseline to week 12 (end of treatment) by:

   i) Reduction in inflammatory and non-inflammatory lesion count ii) IGA success
3. Improvement in patient reported quality of life score using the Skindex-16 questionnaire in participants with acne vulgaris from baseline to week 12

1.2. Secondary Objectives 1. To evaluate the efficacy of B244 in participants with mild to moderate acne vulgaris from baseline to weeks 2, 4, 8, and 16: i) Reduction in inflammatory and non-inflammatory lesion count ii) IGA success iii) Improvement in patient reported quality of life score using the Skindex-16 questionnaire

1.3. Exploratory Objective

1. To evaluate facial skin microbiota in participants with acne vulgaris at baseline, week 4, week 8, week 12, and week 16 in B244-treated participants compared to placebo from: i) Skin swabs will be taken from forehead, nose, both cheeks and chin All participants (placebo and B244) will undergo skin swabs and testing.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for enrollment in the study must meet all the following criteria:

1. Male and females age 18 or older
2. Clinical diagnosis of mild to moderate facial acne vulgaris defined as:

   1. ≥5 inflammatory lesions, and;
   2. ≥10 non-inflammatory lesions, and;
   3. IGA 2-3
3. Willing to refrain from using any treatments, other than the investigational product, for acne present on the face. This includes the use of antibiotics for the treatment of acne. Topical acne treatments that do not have significant or measurable systemic absorption (e.g., benzoyl peroxide, salicylic acid) are allowed for treatment of non-facial acne.
4. Willing and able to provide informed consent and to comply with the study protocol.

Exclusion Criteria:

1. Pregnant and/or lactating females
2. Continuous or planned use of tanning booths or excessive sun exposure, in the opinion of the Investigator.
3. Active cystic acne or acne conglobata, acne fulminans, and secondary acne
4. Two or more active nodular lesions
5. Treatment with over-the-counter topical medications for the treatment of acne vulgaris including benzoyl peroxide, topical anti-inflammatory medications, corticosteroids, α-hydroxy/glycolic acid, or topical probiotics including commercially available product AO+Mist on the face within 7 days prior to baseline.
6. Treatment with systemic corticosteroids within 28 days prior to baseline.
7. Treatment with systemic antibiotics or systemic anti-acne drugs within 7 days prior to baseline.
8. Prescription topical retinoid use on the face within 7 days of baseline (e.g., tretinoin, tazarotene, adapalene).
9. Commencement of new hormonal therapy or dose change to hormonal therapy within 90 days prior to baseline. Dose and frequency of use of any hormonal therapy started more than 90 days prior to baseline must remain unchanged throughout the study. Hormonal therapies include, but are not limited to, estrogenic and progestational agents such as birth control pills.
10. Use of androgen receptor blockers (such as spironolactone or flutamide) in the 7 days prior to randomization.
11. Oral retinoid use (e.g., isotretinoin) within 180 days prior to baseline or vitamin A supplements greater than 10,000 units/day within 180 days of baseline.
12. Cosmetic facial procedures (chemical or laser peel, microdermabrasion, etc.) within the 28 days of the first dose or during the study.
13. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
14. Any condition that the study Investigator feels would indicate that participation would not be in the best interest of the participant.
15. The participant has been previously randomized in this study.
16. The participant has received an investigational product within 30 days or 5 half-lives, whichever is longer prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah Craft, MD, Principal Investigator — Science 37
Locations (1):
- Science37, Culver City, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- B244 Arm: B244 dose (4x10E9 cells/mL) administered in a 1:1 (active vs placebo) ratio
  B244: 4 pumps of spray to saturate the entire face applied BID. Applications should occur in the morning and at night for 12 weeks.
Period: Overall Study
Arm/Group | B244 Arm | Placebo Arm
Started | 186 | 186
Completed | 152 | 148
Not Completed | 34 | 38
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 5 | 7
Not completed — Lost to Follow-up | 15 | 8
Not completed — Withdrawal by Subject | 10 | 21
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: Efficacy analysis set: all subjects who received at least 1 application of IP
Groups:
- Total: Total of all reporting groups
Arm/Group | B244 Arm | Placebo Arm | Total
Number analyzed (Participants) | 181 | 179 | 360
Age, Customized [Count of Participants; unit: Participants]
  18 to <30 years | 126 | 122 | 248
  30 to <65 years | 55 | 57 | 112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 92 | 187
  Male | 86 | 87 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 37 | 76
  Not Hispanic or Latino | 137 | 141 | 278
  Unknown or Not Reported | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 21 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 9 | 28
  White | 107 | 133 | 240
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 28 | 16 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment RelatedAdverse Events
Description: Safety and tolerability endpoints will consist of all treatment related adverse events reporting during the study duration.
Time Frame: 16 weeks
Population: Efficacy analysis set: all subjects who received at least 1 application of IP
Measure: Count of Participants; unit: Participants
Arm/Group | B244 Arm | Placebo Arm
Number analyzed (Participants) | 181 | 179
Participants
  At Least 1 Treatment Related TEAE | 10 | 9
  At Least 1 Treatment Related SAE | 0 | 0

2. Primary Outcome: Change in Inflammatory and Non-inflammatory Lesion Count
Description: Lesion counting was performed using the digital photos taken by participants and stored inside the study mobile platform by trained personnel only. Every effort was made to have the counting and clinical evaluation done by the same evaluator for a given participant. Lesions under the jaw line or behind the hairline (including eyebrows) were not included in the counts. Papules, pustules, cysts and nodules were classified as inflammatory acne lesions, and open and closed comedones were classified as non-inflammatory lesions.
Time Frame: 12 weeks
Population: Efficacy analysis set: all subjects who received at least 1 application of IP
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | B244 Arm | Placebo Arm
Number analyzed (Participants) | 181 | 179
lesions
  Change in Inflammatory Lesion Count from Baseline to Week 12 | -4.8 (10.1) | -3.9 (9.13)
  Change in Non-Inflammatory Lesion Count from Baseline to Week 12 | -4.0 (22.0) | -4.9 (20.9)

3. Primary Outcome: Number of Participants Demonstrating Efficacy Measured by Investigator Global Assessment Success
Description: IGA (Investigator's Global Assessment) was used to assess the overall diseases severity on a scale of 0 to 4 (0=clear, 1=almost clear, 2=mild disease, 3=moderate disease, and 4=severe disease). IGA success was defined as a post-baseline score of 0 or 1 (yes=success, no=no success).
Time Frame: 12 weeks
Population: Efficacy analysis set: all subjects who received at least 1 application of IP
Measure: Count of Participants; unit: Participants
Arm/Group | B244 Arm | Placebo Arm
Number analyzed (Participants) | 181 | 179
Participants
  Yes | 25 | 12
  No | 127 | 137
Statistical Analysis 1: Comparison: B244 Arm vs Placebo Arm; Test type: Equivalence — Primary efficacy power calculations assume a >25% difference between B244 treatment and placebo and a 15% dropout. Each of the endpoints comprising the co-primary endpoint will be tested at an alpha level of p<0.05. In order to achieve 90% power with a 5% Type I error rate, a total of 372 participants is required; p = 0.034, ANCOVA

4. Secondary Outcome: Change in Inflammatory and Non-inflammatory Lesion Count by Week
Description: as for outcome 2
Time Frame: Baseline to weeks 2, 4, 8, 12 and 16
Population: Efficacy analysis set: all subjects who received at least 1 application of IP
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | B244 Arm | Placebo Arm
Number analyzed (Participants) | 181 | 179
lesions
  Change in Inflammatory Lesion Count from Baseline to Week 2: number analyzed (Participants) | 173 | 169
  Change in Inflammatory Lesion Count from Baseline to Week 2 | -1.5 (10.9) | -1.3 (9.94)
  Change in Inflammatory Lesion Count from Baseline to Week 4: number analyzed (Participants) | 167 | 166
  Change in Inflammatory Lesion Count from Baseline to Week 4 | -0.8 (10.46) | -0.8 (9.49)
  Change in Inflammatory Lesion Count from Baseline to Week 8: number analyzed (Participants) | 159 | 160
  Change in Inflammatory Lesion Count from Baseline to Week 8 | -3.3 (9.94) | -3.1 (8.75)
  Change in Inflammatory Lesion Count from Baseline to Week 12: number analyzed (Participants) | 151 | 149
  Change in Inflammatory Lesion Count from Baseline to Week 12 | -4.8 (10.1) | -3.9 (9.13)
  Change in Inflammatory Lesion Count from Baseline to Week 16: number analyzed (Participants) | 151 | 148
  Change in Inflammatory Lesion Count from Baseline to Week 16 | -3.2 (20.6) | -4.0 (11.4)
  Change in Non-Inflammatory Lesion Count from Baseline to Week 2: number analyzed (Participants) | 173 | 169
  Change in Non-Inflammatory Lesion Count from Baseline to Week 2 | -0.9 (17.1) | -2.1 (18.4)
  Change in Non-Inflammatory Lesion Count from Baseline to Week 4: number analyzed (Participants) | 167 | 166
  Change in Non-Inflammatory Lesion Count from Baseline to Week 4 | -1.5 (21.3) | -4.6 (19.1)
  Change in Non-Inflammatory Lesion Count from Baseline to Week 8: number analyzed (Participants) | 159 | 160
  Change in Non-Inflammatory Lesion Count from Baseline to Week 8 | -4.1 (20.4) | -5.8 (17.4)
  Change in Non-Inflammatory Lesion Count from Baseline to Week 12: number analyzed (Participants) | 151 | 149
  Change in Non-Inflammatory Lesion Count from Baseline to Week 12 | -4.0 (22.0) | -4.9 (20.9)
  Change in Non-Inflammatory Lesion Count from Baseline to Week 16: number analyzed (Participants) | 151 | 148
  Change in Non-Inflammatory Lesion Count from Baseline to Week 16 | -6.4 (23.2) | -6.1 (21.7)

5. Secondary Outcome: Number of Participants Demonstrating Efficacy Measured Investigator Global Assessment Score by Week
Description: as for outcome 3
Time Frame: Baseline to weeks 2, 4, 8, 12 and 16
Population: Subjects from the efficacy analysis set (all subjects who received at least 1 application of IP) that remained in the study up to each respective time point for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | B244 Arm | Placebo Arm
Number analyzed (Participants) | 181 | 179
Participants
  Week 2: number analyzed (Participants) | 174 | 170
  Week 2: Yes | 12 | 13
  Week 2: No | 162 | 157
  Week 4: number analyzed (Participants) | 168 | 166
  Week 4: Yes | 9 | 13
  Week 4: No | 159 | 153
  Week 8: number analyzed (Participants) | 160 | 160
  Week 8: Yes | 16 | 10
  Week 8: No | 144 | 150
  Week 12: number analyzed (Participants) | 152 | 149
  Week 12: Yes | 25 | 12
  Week 12: No | 127 | 137
  Week 16: number analyzed (Participants) | 152 | 148
  Week 16: Yes | 12 | 17
  Week 16: No | 140 | 131

6. Secondary Outcome: Change in Patient Reported Quality of Life Score Using the Skindex-16 Questionnaire
Description: The Skindex 16 questionnaire was assigned to subjects to examine the relationship between the subject's skin health and quality of life. Subjects scored 16 questions from 0 to 6 (0=never bothered, 6=always bothered). Total scores could range between 0 to 96, where a higher score is associated with a worse quality of life.
Time Frame: Baseline to weeks 2, 4, 8, 12 and 16
Population: Efficacy analysis set: all subjects who received at least 1 application of IP
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B244 Arm | Placebo Arm
Number analyzed (Participants) | 181 | 179
score on a scale
  Change from Baseline to Week 2: number analyzed (Participants) | 178 | 174
  Change from Baseline to Week 2 | -0.6 (1.05) | -1.6 (0.97)
  Change from Baseline to Week 4: number analyzed (Participants) | 169 | 171
  Change from Baseline to Week 4 | -0.7 (1.10) | -0.7 (1.12)
  Change from Baseline to Week 8: number analyzed (Participants) | 164 | 160
  Change from Baseline to Week 8 | -0.6 (1.23) | -0.7 (1.16)
  Change from Baseline to Week 12: number analyzed (Participants) | 153 | 151
  Change from Baseline to Week 12 | -0.7 (1.16) | -0.6 (1.17)
  Change from Baseline to Week 16: number analyzed (Participants) | 152 | 148
  Change from Baseline to Week 16 | -0.8 (1.16) | -0.7 (1.17)

7. Other Pre Specified Outcome: To Evaluate Facial Skin Microbiota
Description: Evaluate if B244 administration on skin twice daily will affect the microbial content on collected skin swab samples.
Time Frame: baseline, week 4, week 8, week 12, and week 16
Population: Data was not collected for this exploratory endpoint.
Arm/Group | B244 Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 16.
Description: Participants will report adverse events immediately to the Investigator and study personnel. Participants will also be solicited for adverse events at each scheduled visit. Limited vital signs may be measured at home intermittently and recorded in the study mobile application by the participants.
Arm/Group | B244 Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/181 | 0/179
Serious Adverse Events (participants affected / at risk) | 3/181 | 2/179
Other Adverse Events (participants affected / at risk) | 39/181 | 42/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B244 Arm (N=181) | Placebo Arm (N=179)
Pyrexia (General disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B244 Arm (N=181) | Placebo Arm (N=179)
Blepharitis (Ear and labyrinth disorders) | 1 | 0
Ear disorder (Eye disorders) | 1 | 0
Eyelid irritation (Ear and labyrinth disorders) | 0 | 1
Eczema eyelids (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Carbuncle (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Conjunctivitis bacterial (Gastrointestinal disorders) | 1 | 0
Folliculitis (Gastrointestinal disorders) | 1 | 0
Kidney infection (Gastrointestinal disorders) | 1 | 0
Localised infection (Gastrointestinal disorders) | 1 | 0
Nasopharyngitis (Gastrointestinal disorders) | 1 | 0
Sycosis barbae (Gastrointestinal disorders) | 1 | 0
Concussion (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Post-traumatic neck syndrome (General disorders) | 1 | 0
Ulcer (General disorders) | 0 | 1
Xerosis (General disorders) | 1 | 1
Arthralgia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Back pain (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 1 | 1
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 0 | 2
Sexually transmitted disease (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 2 | 2
Tinea blanca (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Viral infection (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 7 | 6
Sunburn (Injury, poisoning and procedural complications) | 0 | 1
Psychiatric disorders (Investigations) | 3 | 0
Blood pressure increased (Investigations) | 0 | 1
Depression (Investigations) | 3 | 0
Panic attack (Investigations) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1
Allergic sinusitis (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dyspnoea (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash pruritic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Hypertension (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may not publish or otherwise publicly disclose the analyzed study data and conclusions drawn from the study without the written consent of Sponsor.

DOCUMENTS (2):
  • Study Protocol (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT02832063/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT02832063/SAP_001.pdf